CLINICAL TRIAL: NCT02259959
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Inhalative Doses (2 μg/5 μg, 10 μg/5 μg, and 40 μg/10 μg) of BI 1744 CL in Fixed Dose Combination With Tiotropium Bromide for 14 Days in Healthy Male Volunteers (Double-blind, Randomised, Placebo Controlled [at Each Dose Level] Study)
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Inhalative Doses of BI 1744 CL in Fixed Dose Combination With Tiotropium Bromide in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.2
Record Dates: First submitted 2014-10-07; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Solutions; Inhalation; Tiotropium Bromide

ARMS (2):
- BI 1744 CL in combination with Tiotropium (Experimental)
  Interventions: Drug: Single rising doses of BI 1744 CL, solution for oral inhalation; Drug: Tiotropium, fixed dose, solution for oral inhalation
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Single rising doses of BI 1744 CL, solution for oral inhalation
  Arms: BI 1744 CL in combination with Tiotropium
Drug: Tiotropium, fixed dose, solution for oral inhalation
  Arms: BI 1744 CL in combination with Tiotropium
Drug: Placebo
  Arms: Placebo

SUMMARY:
To investigate safety, tolerability, pharmacokinetics and pharmacodynamics of BI 1744 CL and Tiotropium Bromide when given as fixed dose combination

ELIGIBILITY:
Inclusion Criteria:

* Healthy male based upon a complete medical history, including physical examination, regarding vital signs (BP, PR), 12-lead ECG measurement, and clinical laboratory tests. There is no finding deviating from normal and of clinical relevance. There is no evidence of a clinically relevant concomitant disease
* Age ≥21 and ≤45 years
* BMI ≥18.5 and <30 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with good clinical practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR, and ECG measurements) deviating from normal and of clinical relevance
* Evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to the drug or its excipients) as judged clinically relevant by the investigator
* Intake of drugs with a long half-life (>24 hours) within at least 1 month or less than 10 half-lives of the respective drug prior to randomization
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to randomisation
* Participation in another trial with an investigational drug within 2 months prior to randomisation
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days as judged by the investigator
* Alcohol abuse (more than 40 g alcohol a day)
* Drug abuse
* Blood donation (more than 100 mL blood within 4 weeks prior to randomisation or during the trial)
* Excessive physical activities within 1 week prior to randomisation or during the trial
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of the study centre

The following exclusion criteria are specific for this study due to the known class side effect profile of ß2-mimetics:

* Asthma or history of pulmonary hyperreactivity
* Hyperthyrosis
* Allergic rhinitis in need of treatment
* Clinically relevant cardiac arrhythmia
* Paroxysmal tachycardia (>100 beats per minute)

The following exclusion criteria are specific for this study due to the known class side effect profile of Tiotropium:

* Hypersensitivity to tiotropium and/or related drugs of these classes
* History of narrow-angle glaucoma
* History of prostatic hyperplasia
* History of bladder-neck obstruction

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-04; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with clinically relevant findings in physical examination | Up to day 32
Number of subjects with clinically relevant findings in vital signs | Up to day 32
  blood pressure, pulse rate
Number of subjects with clinically relevant findings in 12-lead ECG | Up to day 32
Number of subjects with clinically relevant findings in laboratory tests | Up to day 32
Number of subjects witch clinically relevant changes in additional safety laboratory test parameters | up to 318 hours after start of treatment
  Systemic metabolic parameters: cyclic adenosine mono phosphate (cAMP) and potassium
Number of subjects with clinically relevant changes in airway resistance (Raw) measured by body plethysmography | Pre-dose, up to 408 hours after start of treatment
Number of subjects with adverse events | Up to day 32
Global assessment of tolerability by investigator on a 4-point scale | Up to day 32

SECONDARY OUTCOMES:
Maximum concentration in plasma (Cmax) | up to 504 hours after start of treatment
Time from dosing to maximum concentration in plasma (tmax) | up to 504 hours after start of treatment
Area under the concentration-time curve in plasma (AUC) | up to 504 hours after start of treatment
Area under the concentration-time curve in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 504 hours after start of treatment
Percentage of AUC 0-∞ that is obtained by extrapolation (%AUCtz-∞) | up to 504 hours after start of treatment
Terminal rate constant in plasma (λz) | up to 504 hours after start of treatment
Terminal half-life in plasma (t½) | up to 504 hours after start of treatment
Mean residence time in the body after inhalation (MRTih) | up to 504 hours after start of treatment
Apparent clearance after extravascular administration (CL/F) | up to 504 hours after start of treatment
Apparent volume of distribution during the terminal phase λz following an extravascular dose (Vz/F) | up to 504 hours after start of treatment
Amount eliminated in urine from the time point t1 to t2 (Aet1-t2) | up to 336 hours after start of treatment
Fraction excreted in urine from time point t1 to t2 (fet1-t2) | up to 336 hours after start of treatment
Renal clearance from the time point t1 until the time point t2 (CLR,t1-t2) | up to 504 hours after start of treatment
Minimum measured concentration in plasma at steady state over a uniform dosing interval τ (Cmin,ss) | up to 504 hours after start of treatment
Predose concentration of the analytes in plasma at steady state immediately before administration of the next dose (Cpre,ss) | Pre-dose every 24 hours
Time of last measurable concentration in plasma (tz) | up to 504 hours after start of treatment
Linearity index (LI) | up to 504 hours after start of treatment
Accumulation ratio based on Cmax (RA,Cmax) | up to 504 hours after start of treatment
Accumulation ratio based on AUCτ (RA,AUC) | up to 504 hours after start of treatment